CLINICAL TRIAL: NCT06787989
Title: Treatment of Refractory Immune Thrombocytopenia
Brief Title: BCMA-CD19 CCAR T Cell Treatment of Refractory Immune Thrombocytopenia Associated with Autoimmune Diseases
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: iCell Gene Therapeutics (Industry)
Collaborators: iCell ImmunityX（Hangzhou）Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ICG318-ITP-01
Record Dates: First submitted 2025-01-08; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Refractory Immune Cytopenia
Keywords: immune thrombocytopenia; CAR T cells; BCMA-CD19 cCAR; autoimmune diseaases
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BCMA-CD19 cCAR T cells (Experimental): Dose escalation phase: patient's T cells will be transduced with a retroviral vector to express a BCMA-CD19 cCAR. with an escalation approach.
  Interventions: Biological: BCMA-CD19 cCAR T cells

INTERVENTIONS:
Biological: BCMA-CD19 cCAR T cells — • BCMA-CD19 cCAR T cells are used to treat patients. Patient will be administered either fresh or thawed CAR T cells by IV injection after receiving lymphodepleting chemotherapy.

SUMMARY:
This is a phase I, interventional, single arm, open label, treatment study to evaluate the safety and tolerability of BCMA-CD19 cCAR T cells in patients with refractory ITP associated with autoimmune disease.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) Can be associated with various autoimmune diseases, including SLE, and SS. Patients with refractory thrombocytopenia often have long hospital stays, high medical costs, high demand for blood products, and are prone to complications of other systemic injuries. Such patients require active treatment to reduce the risk of life-threatening bleeding, delay the progression of the disease prognosis Glucocorticoids combined with immunosuppressive agents are still the main treatment strategies. Recently, biological agents targeting abnormal immune cells, such as rituximab and belimumab, which deplete B cells have also achieved some success in the treatment of ITP. However, these agents cannot permanently reverse the production of abnormal antibodies as they are unable to eliminate pathogenic long-lived plasma cells because these agents cannot penetrate lymph nodes and soft tissue. The BCMA-CD19 cCAR T-cells are designed to deplete antibody-producing 'root", B cells and plasma cells.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18~60 years old; 2. Diagnosed with immune thrombocytopenia associated with autoimmune diseases including systemic lupus erythematosus (according to the 1997 or 2009 ACR classification criteria), primary Sjogren's syndrome (according to the 2002 ACR/EULAR international classification criteria), undifferentiated connective tissue disease (according to the 1999 international classification criteria). Or patient without clinical manifestations related to connective tissue disease, but with positive anti nuclear antibodies (≥ 1:100) and/or without positive anti SSA/Ro-52 antibodies;Serum creatinine <221.0μmol/L (2.5mg/dl); 3. platelet count<30 × 10 ⁹/L or platelet count ≥ 20 × 10 ⁹/L, accompanied by bleeding symptoms (bleeding symptom score ≥ 2 points). No obvious active infection; 4. Voluntary participation and informed consent signed by the patient or his/her legal/authorized representative.

Exclusion Criteria:

- 1. Serious accompanying diseases that researchers consider clinically significant due to poor control, such as (but not limited to) neurological, cardiovascular, renal, liver, endocrine, or gastrointestinal diseases CNS disease: Active central nervous system (CNS) lupus (including epilepsy, psychosis, organic encephalopathy syndrome, cerebrovascular accident [CVA], encephalitis or CNS vasculitis), visual Disorders, cranial neuropathy requiring intervention 2. Abnormal liver function: aspartate transaminase (AST) or alanine transaminase (ALT) or glutamyl transpeptidase (GGT) detection value is greater than 1.5 times the upper limit of normal (ULN);; urinary protein quantification>1g/24h.

3. History of malignant tumors 4. Active hepatitis B or C.，and HIV positive 5. Individuals with a history of drug allergies or allergies. 6. Have any other clinically significant disease history or current disease that, in the judgment of the research physician, may pose a risk to the safety of the subjects, or interfere with the completion of the research procedure and the evaluation of safety and efficacy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-31 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
The number and incidence of adverse events after BCMA-CD19 cCAR T cell infusion | 24 months
  Evaluation all possible adverse reactions, including the number, incidence, and severity of symptoms such as cytokine release syndromes and neurotoxicity within 3 months after BCMA-CD19 cCAR infusion.

SECONDARY OUTCOMES:
Overall remission rate 12 weeks after BCMA-CD19 cCAR | 24 months
  1. Complete response (CR): Platelet count ≥ 100 × 109/L and no bleeding;
  2. Partial response (PR): platelet count<100 × 109/L, but increased by at least 2 times compared to baseline platelet count, with no bleeding symptoms
  3. Disease control: Disease control monitored up to 2 years after BCMA-CD19 cCAR T cells infusion)

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No